CLINICAL TRIAL: NCT05612113
Title: Live Supervision in Psychotherapy: Study Protocol for a Single Case Experimental Design Study (SCED) With Multiple Baselines in an Outpatient Clinical Setting
Brief Title: Live Supervision in Psychotherapy: Study Protocol for a Single Case Experimental Design Study (SCED)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sven Alfonsson, PhD, Karolinska Institutet
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 2022-00352-01
Record Dates: First submitted 2022-10-17; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Competence
Keywords: Clinical Supervision; Therapist Competence; Training and Supervision; Live Supervision; Psychotherapy; Bug-in-the-Ear

STUDY DESIGN:
Intervention Model Description: Replicated Single Case Experimental Design with Multiple Baselines
Who Masked: Outcomes Assessor
Masking Description: Third-party raters, not being involved in the project management of the study or participating in the study, will be blinded to the participating therapists, study phases and the order of recorded sessions. These third-party raters will assess therapists' skills, goal attainment and competences in each recorded session. To test for blinding integrity the third-party raters will note their guesses of which condition the session belonged to (baseline or intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline - Session Goal Formulation (Active Comparator): In the baseline phase, the therapist will formulate two session goals, see under descriptions of primary outcome measure.
  In this SCED-study, the baseline phase will be of randomized length (5-9 sessions) for each therapist.
  The reason for defining this as an active comparator is that we the behavior of formulating two session goals before each session should be considered an intervention, stimulating the therapist to reflect on the upcoming session goals, on defining concrete behaviors to reach the session goal, and to reflect upon his/her session behaviors afterwards. Thus, regarding the baselinephase as a no intervention would be misleading.
  Interventions: Other: Session Goal Formulation
- Live Supervision with Bug-in-the-Ear (BITEar) as method (Experimental): LS with the Bug-in-the-Ear (BITEar) is a video based supervision format where the supervisor watches the therapy session live through a webcam in the therapy room. During the therapy session, the supervisor provide verbal feedback and guidance to the therapist who wears wireless in-ear headphones.
  In this SCED-study, the intervention phase consist of 5 to 9 BITEar supervision sessions (number of supervision sessions is randomized between therapists)
  The BITEar supervision will consist of three phases:
  Pre-supervision (15 minutes): Discussion of the therapists session goals, how the therapist wants the supervisor's help and agreement on prompts and cues from supervisor
  Live supervision during the therapy session (≈ 45-60 minutes): Supervisor gives real time feedback and guidance focusing on helping the therapist achieve session goals
  Post-supervision (15 minutes): Reflection about the session, session goals and the supervision.
  Interventions: Behavioral: Live Supervision + Session Goal Formulation

INTERVENTIONS:
Behavioral: Live Supervision + Session Goal Formulation — Read under "Arms"
  Arms: Live Supervision with Bug-in-the-Ear (BITEar) as method
Other: Session Goal Formulation — Read under "Arms"
  Arms: Baseline - Session Goal Formulation

SUMMARY:
Although clinical supervision is an essential part of psychotherapy training and development, the empirical evidence for effects on therapist competence and patient outcome is limited. However, a novel format, Live Supervision (LS), enables real time feedback during the patient session which counteracts on several of the major identified problems with standard supervision. Pilot studies of LS show promising results, but the effects of LS has never been assessed in a clinical setting with licensed psychologists. Furthermore, manualized LS with a stringent focus at therapists' idiosyncratic challenges has never been evaluated.

The primary aim of this study is to evaluate the effects of LS on therapist competence and perceived therapy challenges in a clinical outpatient setting with licensed psychologists as therapists. Secondary aims are to examine when and how LS is optimal for clinical supervision.

DETAILED DESCRIPTION:
Objective:

To evaluate the effects of LS on therapist competence and perceived therapy challenges with both qualitative and quantitative data in a sample of licensed psychotherapists working with CBT in outpatient psychiatry or primary care.

Methods:

The study will use a replicated Single Case Experimental Design (SCED) with randomized multiple baselines in combination with qualitative interviews at the end of the trial. Each therapist (n = 6) will take part in the study with one patient for a period of 14 therapy sessions of which 5-9 sessions (randomized for each therapist) consist of the baseline phase, followed by the intervention phase (Live Supervision) for the rest of the study period (5-9 sessions).

Primary outcome measures will be observer rated competence and observer and therapist rated goal attainment. Secondary outcome measure will be the quality of therapy sessions from the perspective of the patients and observer rated competence according to the supervisors perception of the most prevalent skill deficiency of the therapist.

The qualitative data collection will focus on a systemization of how and when LS is for optimal use as well as mapping the degree of correspondence between patients, therapists, and supervisors regarding the therapists competences and skill deficiencies.

ELIGIBILITY:
Patients:

Inclusion Criteria:

1. At least one diagnosis of the following DSM-5 disorders: mood disorders, anxiety disorders, OCD or related disorders, orTrauma or stress related disorders, comorbid severe disorder such as schizophrenia or development disorder,
2. Being able to attend to regular treatment
3. Accepting recording of therapy sessions and providing a written consent
4. Above 16 years old

Exclusion Criteria:

a) Comorbid severe disorder such as schizophrenia, developmental disorder, severe eating disorder, or severe substance use disorder.

Therapists:

Inclusion criteria:

1. Licensed psychologist
2. Working in outpatient psychiatric care or primary care in Sweden
3. Currently providing CBT
4. At least one year work experience of providing psychological treatments in outpatient care

Supervisors:

Inclusion criteria:

1. At least 2 years experience working as a clinical supervisor for CBT
2. Formal supervision training

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Therapist Rated Session Goal Attainment of Idiosyncratically Formulated Session Goals | Approximately 14 weeks (from session 1 to session 14 with one session per week)
  All therapists will formulate two individual development goals per therapy session for the 14 weeks. One goal is focusing on a challenging behavioral pattern of the patient (e.g. talkative), and the other focusing on a challenging behavior of the therapist (e.g. being concise).
  After each session, each therapist rates to what degree they perceived that they managed to reach each of their set up goals on a scale from 0 (not reached the goal at all) to 100 (fully reached the goal) with 5 anchor points with descriptions. They will also rate the perceived difficulty of working with the goal from a scale from 0 (not at all difficult) to 100 (extremely difficult) with 5 anchor points with descriptions.
Observer Rated Session Goal Attainment of Idiosyncratically Formulated Session Goals | Approximately 14 weeks (from session 1 to session 14 with one session per week)
  Third-party raters will listen to the audio recordings of the sessions and evaluate the level of goal attainment in each session, blinded to whether the therapist received supervision or not. Observers will be trained in how to evaluate goal attainment.
Therapist Competence measured with Cognitive Therapy Scale - Revised (CTS-R; Blackburn et al., 2001) | Approximately 14 weeks (from session 1 to session 14 with one session per week)
  The CTS-R instrument is one of the most used and validated scales for measuring CBT competence. The scale consists of 12 items with a 7-point rating scale format: 0 = poor, 1 = barely adequate, 2 = mediocre, 3 = satisfactory, 4 = good, 5 = very good, and 6 = excellent.
  In this study, we will analyze both the composite score of the full scale, but also an item per item analysis since one of the aims of the study is to assess for what type of competencies LS may be particularly effective.

SECONDARY OUTCOMES:
Patient rated degree of satisfaction and usefulness | Approximately 14 weeks (from session 1 to session 14 with one session per week)
  Each session, the patient will rate how satisfied and how useful they perceived the session. The rating is on a scale from 0 (not at all) to 100 (extremely)
Patient rated degree of collaboration with the therapist | Approximately 14 weeks (from session 1 to session 14 with one session per week)
  As a proxy measure for therapeutic alliance, a single item will be used where the patient is asked to rate how they perceived the collaboration with their therapist on a scale from 0 (not good at all) to 100 (extremely good).
Observer rated degree of therapist skill deficiency as defined by the supervisor | Approximately 14 weeks (from session 1 to session 14 with one session per week)
  During the interviews in the end of the trial, the supervisors will be asked to define the most important therapist skill deficiency. This skill will then be operationalized and rated for each session by a blinded third party rater.
Observer rated degree of therapist skill deficiency as defined by the patient | Approximately 14 weeks (from session 1 to session 14 with one session per week)
  During the interviews in the end of the trial, the patients will be asked to define the most important therapist skill deficiency. This skill will then be operationalized and rated for each session by a blinded third party rater.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Alfonsson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institute, Stockholm, Region Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No